CLINICAL TRIAL: NCT03833622
Title: Shared Decision Making to Improve Goals of Care Discussions in the Emergency Department
Brief Title: Shared Decision Making to Improve Goals of Care in the ED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Laura E. Walker, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-000128
Record Dates: First submitted 2018-01-03; First posted 2019-02-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Goals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shared decision aid assessment (Experimental): Patients will be selected to have a goals of care discussion with an emergency physician utilizing a pilot decision aid and will be asked for feedback to assist with refinement of the decision aid.
  Interventions: Other: Shared Decision Aid Assessment

INTERVENTIONS:
Other: Shared Decision Aid Assessment — Provide feedback on a shared decision making tool to aid in discussion on goals of care in the emergency department

SUMMARY:
This project will develop and refine a shared decision making (SDM) intervention (decision aid tool) to improve and normalize high quality end of life discussions in the Emergency Department (ED) setting.

DETAILED DESCRIPTION:
Develop a shared decision making (SDM) intervention informed by insights elicited from patients and clinicians to improve goals of care discussions.

The process of decision aid design involves: (1) review and synthesis of the evidence; (2) an analysis of usual practice through observation of clinical encounters; (3) development of an initial decision aid prototype; (4) field testing in the context of clinical care to gain insights on both intended and unintended effects of its use in practice to facilitate patient centered goals of care discussions; and (5) successive iterations of the decision aid until thematic saturation is reached and it is ready for testing in a clinical trial.

ELIGIBILITY:
Inclusion:

1. Patients presenting to Mayo Clinic Rochester, Saint Marys' Emergency Department,
2. Patients at high risk for critical illness as determined by an Elderly Risk Assessment (ERA) score ≥ 16 or as determined by provider discretion,
3. ≥ 60 years of age,
4. Ability to provide informed consent,
5. Medically stable at the time of enrollment,
6. Able to participate without causing a delay in care.

Exclusion:

1. GCS scores < 15,
2. Signs of altered mental status,
3. Known to be pregnant,
4. Incarcerated or in Police Custody,
5. Communication barriers such as visual or hearing impairment that may preclude use of the decision aid.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient and physician feedback survey for tool development and iterative refinement | 1 year
  A debrief survey/open-ended questionnaire is filled out by the patient and his/her provider to collect feedback. This is used to refine this shared decision making (SDM) intervention in the Emergency Department (ED) setting.

SECONDARY OUTCOMES:
Patient and physician satisfaction questionnaire | 1 year
  A satisfaction questionnaire is filled out by the patient and his/her provider following conversation on goals of care either with or without the SDM intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Laura E Walker, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials (best in chrome) — https://www.mayo.edu/research/clinical-trials